CLINICAL TRIAL: NCT00897754
Title: Alternative Splice Forms of VEGF in Colorectal Cancer - Possible Value in Anti-VEGF Therapy
Brief Title: Gene Expression in Patients With Advanced or Metastatic Colorectal Cancer Receiving Bevacizumab
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000560986; ECOG-E3200T2
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; stage III colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: immunologic technique

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors understand how patients respond to treatment.

PURPOSE: This laboratory study is looking at gene expression in patients with advanced or metastatic colorectal cancer receiving bevacizumab.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the balance of splice form expression alters susceptibility of tumors in vivo to respond to anti-VEGF therapy.

OUTLINE: Tumor tissue samples collected on clinical trial E-3200 are analyzed for laboratory endpoints.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor tissue samples available from patients with advanced or metastatic adenocarcinoma of the colon or rectum

  * Receiving bevacizumab on clinical trial E-3200

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E3200
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-07-24 (Actual); Primary Completion 2009-02-01 (Actual); Study Completion 2009-02-01 (Actual)

PRIMARY OUTCOMES:
Mean scores for VEGFb and pan-VEGF gene expression by IHC | 1 month
Gene expression as measured by tissue microarrays | 1 month
Splice form expression as measured by reverse transcriptase-PCR | 1 month
VEGF165b protein expression as measured by ELISA | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: David Bates, PhD, Study Chair — Bristol Heart Institute at University of Bristol